CLINICAL TRIAL: NCT05447299
Title: Neurobiomekaniska Modeller av Spasticitet Med hjälp av Personspecifika Muskelparametrar
Brief Title: Neuromusculoskeletal Modeling of Muscle Spasticity
Status: Enrolling by invitation | Type: Observational
Sponsor: Region Stockholm (Other Government)
Collaborators: Karolinska University Hospital (Other); KTH Royal Institute of Technology (Other); Karolinska Institutet (Other)
Responsible Party: Sponsor
Other Study IDs: K 0000-0001
Record Dates: First submitted 2022-06-13; First posted 2022-07-07 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-04

CONDITIONS: Cerebral Palsy; Musculoskeletal Deformity; Spasticity; Muscle Strength; Walking, Difficulty
Keywords: Spastic cerebral palsy; Muscle function; Hyper-resistance; Functional mobility
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity; Mobility Limitation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Typically developing children: Reference group of typically developing children
- Cerebral palsy group: Children with a diagnosis of cerebral palsy

SUMMARY:
Cerebral palsy (CP) is a movement and posture disorder caused by an injury to the developing brain, with a prevalence in Sweden of about 2/1000 live births. Children with CP have walking difficulties, and decreased muscle mass and muscle function as compared to typically developing (TD) children. The extent of disability in CP depends on the severity and timing of the primary cerebral lesion and can be classified with the gross motor function classification system (GMFCS E&R) that ranges from walking without limitations (I) to being transported in a wheelchair (V).

Muscle function commonly deteriorates with age and contracture development is often clinically evident as early as at 4 years of age. In addition to being thinner and weaker, skeletal muscle in children with CP develop poor quality, i.e., increasingly higher amounts of fat and connective tissue at the expense of functional, contractile proteins.

How long-term standard treatments for children with spastic CP including, training and orthotics use, with botulinum toxin (BoNT-A) treatment as an adjunct, affects muscle on functional, structural, and microscopic level in CP has not yet been published. Therefore, we will investigate the muscle function as well as functional mobility, structure, and spasticity. We will conduct functional mobility tests. Muscle strength will be measured with a rig-fixed dynamometer, and muscle structure will be measured with magnetic resonance imaging. The spasticity will be instrumentally assessed by the NeuroflexorTM, a machine measuring resistance in a muscle when a pedal is passively moving the participants foot at two different speeds. We will follow participants, for 1 year, with 4 measurements during this period.

In order to better treat these children, we need to better understand the complex, interrelated interactions of musculoskeletal properties and function in children with CP. Our hypothesis is that muscle structure and function is affected by standard clinical treatments sessions including routine botulinum toxin treatment. Analyzing the effect of standard care may help planning of more effective clinical treatments in the future.

DETAILED DESCRIPTION:
How long-term standard treatments for children with spastic cerebral palsy (CP), including training and orthotics use, with botulinum toxin (BoNT-A) treatment as an adjunct, affects muscle on functional, structural, and microscopic level in CP has not yet been published. Therefore, we will investigate the muscle function as well as functional mobility, structure, and spasticity.

Research questions:

* How is muscle structure, muscle strength, spasticity and, stiffness of the calf muscle in CP related to motor function, and how does it differ to typically developing (TD) children?
* What is the long-term effect of a standard care with BoNT-A as an adjunct on motor function, muscle structure, muscle strength, spasticity, and stiffness?

Participants with spastic CP, aged between 5-17 years, are recruited from the Dept of Pediatric Orthopaedics, when clinically motivated plans for the first BoNT-A treatment session of the calf (plantar flexors) are set. Typically developing children at same ages are recruited through convenient sample and will take part of the assessments once. The children with CP will go through the following assessments at four different time-points; before, 3 months, 6 months, and one year after the first BoNT-A injection:

* Spasticity will be measured with clinical tests: Modified Tardieu scale and Modified Ashworth scale and with a instrumented device measuring muscle resistance, the NeuroflexorTM.
* Isometric strength measurements of plantar flexors and ankle dorsiflexors using a dynamometer (ChatillonTM) fixed in a custom-built testing frame while surface EMG is captured.
* Functional mobility in walking for example the Timed-Up-and-Go test (TUG-test) i.e. the time it takes for the child to stand up from a chair, walk 3 m, turn around, walk back, and sit down.
* Active and passive range of motion (ROM) measured with a goniometer

Before the first injection, the children with CP will be examined with magnetic resonance imaging (MRI) providing complex 3D structural information of individual muscles. One year after first injection, another examination with MRI will be conducted.

This explorative, observational, prospective, long time follow up study will be conducted at the Motion analysis laboratory at Astrid Lindgren's children's hospital and Huddinge Karolinska in collaboration with KTH Royal Institute of Technology.

Parametric and/or non-parametric statistical tests for within and between group comparisons, and correlations will be performed. Based on the pilot data from TD children the CP group and previous literature we need a sample size of 10-15 participants in each group.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral/Bilateral spastic CP without Botulinum toxin injection history
* Understanding study protocol and expressing voluntary consent of the family
* Dorsiflexion to at least a neutral position of the foot

Exclusion Criteria:

* Contraindication to MRI scanning: metal fragments in the body, surgically implanted devices containing metal, severe claustrophobia, or inability to lie down in the MRI scanner, presence of pacemaker or other stimulators, shunts etc.
* Total range of ankle movement less than 35°

Ages: 5 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Participants with spastic CP are recruited from the Dept of Pediatric Orthopaedics, Astrid Lindgren Children's Hospital, Karolinska University Hospital, Stockholm, Sweden. The TD children are recruited from siblings of the participants with CP, and friends and family of the research group.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2019-01-15 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in muscle structure | Before and one year after the first treatment session
  MRI based examinations including muscle volume
Change in spasticity | Before, three months, six months and 12 months after the firstt treatment session
  Resistance at slow and fast passive movements of the foot
Change in muscle strength | Before, three months, six months and 12 months after the first treatment session
  Muscle strength measured as force with a dynamomter in the calf muscle
Change in functional mobility during walking | Before, three months, six months and 12 months after the first treatment session
  Time to complete a test of functional mobility during walking will be measured

CONTACTS AND LOCATIONS:
Overall Officials: R Wang, Ing, PhD, Principal Investigator — KTH Royal Institute of Technology
Locations (1):
- Region Stockholm, Karolinska University Hospital, Stockholm, Sweden

REFERENCES:
- [Derived] Ahblom A, Ponten E, Destro A, Petersson S, von Walden F, Wang R, Lidbeck C. Exploration of the triceps surae muscle in ambulatory children with cerebral palsy using instrumented measurements of stiffness and diffusion tensor magnetic resonance imaging for muscle architecture. BMC Musculoskelet Disord. 2024 Oct 11;25(1):803. doi: 10.1186/s12891-024-07890-4. PMID 39394126